CLINICAL TRIAL: NCT00611858
Title: Phase II Study of Cetuximab, 5-FU and Radiation as Neoadjuvant Therapy for Patients With Locally Advanced Rectal Cancer
Brief Title: Cetuximab, 5-FU and Radiation as Neoadjuvant Therapy for Patients With Locally Advanced Rectal Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other); Brigham and Women's Hospital (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jeffrey A. Meyerhardt, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-297; BMS CA225302
Record Dates: First submitted 2008-01-29; First posted 2008-02-11 (Estimated); Results first posted 2018-11-14 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Rectal Cancer
Keywords: 5-FU; cetuximab; radiation; adenocarcinoma of the rectum; neoadjuvant therapy
MeSH Terms: conditions — Rectal Neoplasms | interventions — Cetuximab; Fluorouracil; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cetuximab, 5-FU and Radiation (Experimental): Cetuximab: Participants first receive cetuximab at the initial dose of 400 mg/m2 intravenously (IV) administered over 120 minutes, followed by weekly infusions at 250 mg/m2 over 60 minutes. Cetuximab is given as single agent during the first 3 weeks on study and then in combination with 5-FU and radiation.
  Radiation: Radiation therapy given as standard of care is initiated after the 3rd dose of cetuximab with a total dose of 50.4 Gray (Gy) in 28 fractions over approximately 5.5 weeks.
  5-FU: Participants receive 5-Fluorouracil (5-FU) continuous infusion through central venous access at 225 mg/m2/day given 7 days a week starting day 1 of radiation (no later than 3 days) and lasting the duration of radiation therapy.
  Duration of neoadjuvant therapy is estimated to be 9 weeks. Surgery follows at week 13-17. Sigmoidoscopy is performed for biopsy prior to the 1st dose and after 3rd dose of cetuximab before the initiation of radiation and/or 5-FU.
  Interventions: Drug: Cetuximab; Drug: 5-Fluorouracil; Radiation: Radiation

INTERVENTIONS:
Drug: Cetuximab
  Other Names: Erbitux
Drug: 5-Fluorouracil
  Other Names: 5-FU
Radiation: Radiation
  Other Names: External Beam Radiation Therapy

SUMMARY:
The standard treatment for rectal cancer is to receive the chemotherapeutic drug 5-fluorouracil (5-FU) with radiation therapy before having surgery to remove the rectal cancer. This is known as neoadjuvant chemoradiotherapy. The purpose of this research study is to determine if Cetuximab improves the benefits of neoadjuvant chemoradiotherapy when given with 5-FU and radiation therapy.

DETAILED DESCRIPTION:
The epidermal growth factor receptor (EGFR) present in normal and tumor cells is involved in signaling pathways affecting cellular growth, differentiation, proliferation and programmed cell death. Overexpression of EGFR has been associated with poorer prognosis in colorectal cancer. Cetuximab targets and blocks EGFR and has been shown to be safe and effective in treating colorectal cancer and head and neck cancers.

The primary hypothesis is that cetuximab in combination with standard 5-FU and radiation as neoadjuvant therapy would improve pathological complete response (pCR) compared to the historical rate (30% versus 10%). The regimen would be considered promising if 5 or more of 25 evaluable participants achieve pCR. The probability of observing this outcome is 0.91 and 0.10 if the true pCR rate is 30% and 10%, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum that begins within 15cm of the anal verge as determined by sigmoidoscopy and/or colonoscopy, with no evidence of distant metastatic disease. A complete colonoscopy to the cecum is recommended prior to initiating protocol therapy.
* Staging with transrectal ultrasound or endorectal coil Magnetic resonance imaging (MRI) to confirm clinical stage of T3 or T4 or lymph node positive rectal adenocarcinoma
* Tumor is K-ras wildtype by method of choice at respective institution (testing codons 12 and 13)
* Performance status: Eastern Cooperative Oncology Group Performance Score (ECOG PS) less than or equal to 2
* 18 years of age or older
* No evidence of metastatic disease by abdominal/pelvic (Computed tomography) CT and chest imaging
* Adequate bone marrow, renal,and hepatic function as outlined in protocol
* All patients will be evaluated by a surgeon and considered a candidate for definitive surgery
* Coumadin or heparin management for line care of other indications is permitted. The International Normalised Ratio (INR) will be monitored weekly in patients taking coumadin.

Exclusion Criteria:

* Prior treatment for this malignancy
* Prior history of pelvic radiation therapy
* Prior history of 5-FU based or EGFR receptor inhibitor therapy
* Prior history of an allergic reaction to a monoclonal antibody
* Uncontrolled serious medical or psychiatric illness
* Significant history of uncontrolled cardiac disease
* Sexually active women of childbearing potential must use an effective method of birth control during the course of the study
* Unwilling to agree to pre and post-cetuximab sigmoidoscopy and biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-05; Primary Completion 2012-12 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Meyerhardt, MD, MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - South Shore Hospital, Weymouth, Massachusetts
  - Vanderbilt Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from May 2008 through July 2012.
Groups:
- Cetuximab With Standard 5-FU and Radiation: Cetuximab: Participants first receive cetuximab at the initial dose of 400 mg/m2 intravenously (IV) administered over 120 minutes, followed by weekly infusions at 250 mg/m2 over 60 minutes. Cetuximab is given as single agent during the first 3 weeks on study and then in combination with 5-FU and radiation.
  Radiation: Radiation therapy given as standard of care is initiated after the 3rd dose of cetuximab with a total dose of 50.4 Gray (Gy) in 28 fractions over approximately 5.5 weeks.
  5-FU: Participants receive 5-Fluorouracil (5-FU) continuous infusion through central venous access at 225 mg/m2/day given 7 days a week starting day 1 of radiation (no later than 3 days) and lasting the duration of radiation therapy.
  Duration of neoadjuvant therapy is estimated to be 9 weeks. Surgery follows at week 13-17. Sigmoidoscopy is performed for biopsy prior to the 1st dose and after 3rd dose of cetuximab before the initiation of radiation and/or 5-FU.
Period: Overall Study
Arm/Group | Cetuximab With Standard 5-FU and Radiation
Started | 13
Completed | 9
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab With Standard 5-FU and Radiation
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 56 [40 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Pathological Complete Response Rate
Description: Pathological complete response (pCR) rate is the percentage of participants who achieve pCR defined as no evidence of tumor cells in the surgical specimen including the lymph nodes (down-staging to pathological T0, N0 after planned neoadjuvant therapy).
Time Frame: Disease is assessed at the time of surgery which in this study cohort occurred up to 24 weeks from date of registration.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cetuximab With Standard 5-FU and Radiation: Determine the pathological complete response rate of cetuximab with standard 5-FU and radiation as neoadjuvant therapy in patients with stage II/III rectal cancer.
Arm/Group | Cetuximab With Standard 5-FU and Radiation
Number analyzed (Participants) | 13
percentage of participants | 30.8 [11.3 to 57.3]

2. Secondary Outcome: Local Recurrence Rate
Description: Local recurrence rate is the percentage of participants experiencing recurrence within the pelvis.
Time Frame: CT scans for surveillance recommended yearly x 3 years from date of surgery with additional scanning at discretion of treating oncologist. Mean follow-up for this study cohort was 4.4 years from study entry, up to 7.9 years.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab With Standard 5-FU and Radiation
Number analyzed (Participants) | 13
percentage of participants | 0.0 [0.0 to 20.6]

3. Secondary Outcome: Complete Resection Rate
Description: Complete resection rate is the percentage of participants having all gross disease removed by the surgeon at the time of operation.
Time Frame: Disease is assessed at the time of surgery which in this study cohort occurred up to 24 weeks from date of registration.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab With Standard 5-FU and Radiation
Number analyzed (Participants) | 13
percentage of participants | 100.0 [79.4 to 100.0]

4. Secondary Outcome: Distant Recurrence Rate
Description: Distant recurrence rate is the percentage of participants experiencing recurrence outside the pelvis.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, 5-FU and Radiation
Number analyzed (Participants) | 13
percentage of participants | 0.0 [0.0 to 20.6]

5. Secondary Outcome: Incidence of Grade 4 Treatment-Related Toxicity
Description: All grade 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on NCI Common Toxicity Criteria for Adverse Events version 3 (CTCAEv3) as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 4 AE of any type during the time of observation.
Time Frame: Disease is assessed through the time of surgery which in this study cohort occurred up to 24 weeks from date of registration.
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab, 5-FU and Radiation
Number analyzed (Participants) | 13
Participants | 3

6. Secondary Outcome: 1-Year Overall Survival Rate
Description: 1-year overall survival is the percentage of participants remaining alive 1 year from study entry.
Time Frame: Mean follow-up for this study cohort was 4.4 years from study entry, up to 7.9 years.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, 5-FU and Radiation
Number analyzed (Participants) | 13
percentage of participants | 100.0 [79.4 to 100.0]

7. Other Pre Specified Outcome: 1-Year Disease-Free Survival Rate
Description: Disease-Free Survival Rate is the percentage of participants remaining alive without disease progression.
Time Frame: as for outcome 2
Population: The analysis dataset is comprised of all enrolled patients.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cetuximab, 5-FU and Radiation
Number analyzed (Participants) | 13
percentage of participants | 100.0 [79.4 to 100.0]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are assessed through the time of surgery which in this study cohort occurred up to 24 weeks from date of registration.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv3. All remaining events regardless of treatment attribution were classified as Other AEs. No further data is available to specify classification of other beyond the general term.
Groups:
- Cetuximab With Standard 5-FU and Radiation: Patients with stage II/III rectal cancer who have received cetuximab with standard 5-FU and radiation as neoadjuvant therapy.
Arm/Group | Cetuximab With Standard 5-FU and Radiation
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 6/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab With Standard 5-FU and Radiation (N=13)
Proctitis (Gastrointestinal disorders) | 1
Rectum, pain (Gastrointestinal disorders) | 1
Cytokine release syndrome (Immune system disorders) | 2
Lymphopenia (Investigations) | 2
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Ulceration (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab With Standard 5-FU and Radiation (N=13)
Hypokalemia (Metabolism and nutrition disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 3
Hearing-other (Ear and labyrinth disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 7
Proctitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Oral cavity, hemorrhage (Gastrointestinal disorders) | 1
Rectum, hemorrhage (Gastrointestinal disorders) | 3
Abdomen, pain (Gastrointestinal disorders) | 2
Rectum, pain (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 8
Fever w/o neutropenia (General disorders) | 1
Edema limb (General disorders) | 1
Pain NOS (General disorders) | 2
Infection Gr0-2 neut, middle ear (Infections and infestations) | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 1
Burn (Injury, poisoning and procedural complications) | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 3
Radiation dermatitis (Injury, poisoning and procedural complications) | 1
Leukocytes (Investigations) | 3
Lymphopenia (Investigations) | 2
Neutrophils (Investigations) | 1
Platelets (Investigations) | 1
Weight loss (Investigations) | 1
Alkaline phosphatase (Investigations) | 2
ALT, SGPT (Investigations) | 3
AST, SGOT (Investigations) | 2
Anorexia (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Bicarbonate (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 6
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Back, pain (Musculoskeletal and connective tissue disorders) | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 2
Taste disturbance (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 2
Neuropathy CN XII tongue (Nervous system disorders) | 2
Neuropathy-sensory (Nervous system disorders) | 2
Head/headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 3
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Nail changes (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 11
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 2
Skin-other (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
This study was terminated early due to weak accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No